CLINICAL TRIAL: NCT03990155
Title: Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease With Extracorporeal Carbon Dioxide Removal Associated With High Flow Nasal Cannula Oxygen Therapy. Pilot Study.
Brief Title: Extra-Corporeal Carbon Dioxide Removal in Exacerbations of Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Policlinico Hospital (Other)
Collaborators: Niguarda Hospital (Other); San Gerardo Hospital (Other); Ospedale San Paolo (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, Professor, Policlinico Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fondazione IRCCS Ca' Granda
Record Dates: First submitted 2019-05-27; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Respiratory Failure With Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HFNCOT+ECCO2R (Experimental): Patients on NIV+ECCO2R who have reached at least for 4 consecutive hours, a RR <25 bpm + pH >7.35 + absence of clinical signs of respiratory distress after treatment with NIV+ECCO2R
  Interventions: Procedure: HFNCOT+ECCO2R

INTERVENTIONS:
Procedure: HFNCOT+ECCO2R — NIV will be discontinued, the ECCO2R setting will be unchanged (both sweep gas flow and blood flow through the artificial lung) and HFNCOT will be started, titrating the fraction of inspired Oxygen (FiO2) to obtain an oxygen saturation at periphery (SpO2) 88-92%; HFNCOT start temperature will be 31°C, the initial flow rate will be 60 L/min.

SUMMARY:
Around 20% of the patients requiring hospitalization for Acute Exacerbation of Chronic Obstructive Pulmonary Disease (AECOPD) develop hypercapnia, which is associated with an increased risk of death. Once Non Invasive Ventilation (NIV) has been initiated, a reduction in Respiratory Rate (RR) and improvement in pH within 4 h predicts NIV success. If pH <7.25 and RR >35 breath per minutes persist, NIV failure is likely. Worsening acidosis, after initial improvement with NIV, is also associated with a worse prognosis. In addition, it has been shown that delaying intubation in patients at high risk for NIV failure has a negative impact on patient survival. Hence, assessing the risk of NIV failure is extremely important. NIV has some limitations: a) intolerance, discomfort and claustrophobia requiring frequent interruptions; b) poor patient-ventilator synchrony, especially in presence of air leaks or high ventilatory requirements. Since removing carbon dioxide by means of an artificial lung reduces the minute ventilation required to maintain an acceptable arterial partial pressure of carbon dioxide (PaCO2), the investigators hypothesize that applying Extra-Corporeal CO2 Removal (ECCO2R) in high-risk AECOPD patients may reduce the incidence of NIV failure and improve patient-ventilator interaction. After the beginning of ECCO2R, NIV could be gradually replaced by High Flow Nasal Cannula Oxygen Therapy (HFNCOT), potentially reducing the risk of ventilator induced lung injury, improving patient's comfort and probably allowing the adoption of a more physiologically "noisy" pattern of spontaneous breathing.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to Emergency or Pulmonology Department, with history of COPD (pulmonary function test available, any Global Obstructive Lung Disease -GOLD- stage), treated with NIV for acute hypercapnic respiratory failure due to AECOPD defined by:

* pH <7.35 + PaCO2 >45 mmHg (acute hypercapnic respiratory failure) or pH <7.35 + PaCO2 > 20% of baseline value (acute on chronic hypercapnic respiratory failure)
* Acute worsening of respiratory symptoms that results in additional therapy
* Respiratory failure not fully explainable with cardiac failure and at high risk for NIV failure, defined by:
* No improvement or worsening of respiratory acidosis (pH <7.35 and PaCO2 >45 mmHg) after 2 hours of NIV + one of the following: RR ≥30 bpm; use of accessory respiratory muscle or paradoxical breathing (Combination criteria for NIV failure) or
* Glasgow Coma Scale ≤ 11 after 2 hours of NIV (Single criteria for NIV failure) or
* Inability to fit mask (facial deformity/intervention/burns) or marked intolerance to interface because of patient's agitation (Single Criteria for NIV failure)

Exclusion Criteria:

* Age >80 years old
* Contraindications to anticoagulation (any of the following: platelet count <30.000/mm3; activated partial thromboplastin time (aPTT) >1,5; stroke or severe head trauma or intracranial arteriovenous malformation or cerebral aneurysm in the previous 3 months; central nervous system mass lesion; history of congenital bleeding diatheses; gastro-intestinal bleeding in the previous 6 weeks; gastro-esophageal varices)
* Cirrhosis
* PaO2/FiO2 ≤ 150 mmHg
* Hemodynamic instability (80-90 mmHg increase or 30-40 mmHg decrease systolic arterial pressure compared to baseline value or need of vasopressors to maintain systolic blood pressure higher than 85 mmHg or electrocardiogram evidence of ischemia/arrhythmias)
* Body Mass Index ≥37
* Impending respiratory arrest
* Catheter access to femoral vein or jugular vein impossible
* Patient moribund, decision to limit therapeutic interventions
* Opposition to participate obtained from the patient or their legally acceptable representative

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Number of partecipants failing HFNCOT+ECCO2R treatment with need of restoring NIV or need of invasive mechanical ventilation | Through study completion, an average of 2 years
  ECCO2R+HFNCOT failure criteria are defined by at least two of the following after at least 1 hour of treatment
  1. Respiratory acidosis (pH <7.35)
  2. RR ≥ 30 bpm
  3. Development of progressive hypoxemia (PaO2/FiO2 < 150)
  4. Paradoxical breathing

SECONDARY OUTCOMES:
Number of partecipants failing NIV+ECCO2R treatment with need of invasive mechanical ventilation | Through study completion, an average of 2 years
  NIV+ECCO2R failure is defined by two of the following occurring for at least 2 hours:
  1. No improvement or worsening of respiratory acidosis (pH <7.35)
  2. RR ≥30 bpm
  3. Development of progressive hypoxemia (PaO2/FiO2 ≤150)
Number of patients treated with ECCO2R reporting one or more side effects due to ECCO2R | Through study completion, an average of 2 years
  1. Bleeding (any bleeding event requiring the administration of 1 U of packed red cells)
  2. Vein perforation at cannula insertion
  3. Hemodynamic instability (80-90 mmHg increase or 30-40 mmHg decrease systolic arterial pressure compared to baseline value or need of vasopressors to maintain systolic blood pressure higher than 85 mmHg or electrocardiogram evidence of ischemia/arrhythmias)
  4. Pneumothorax
  5. Ischemic bowel
  6. Acute kidney failure
  7. Neurological complications (occurrence, after initiation of ECCO2R, of ischemic/hemorrhagic ictus or clinical seizure or cerebral oedema)
  8. Metabolic complications (occurrence, after initiation of ECCO2R of hyperbilirubinemia or glucose≥240 mg/dL)
  9. Thromboembolic complications (occurrence, after initiation of ECCO2R, of deep venous thrombosis, pulmonary embolism)
Variation of pulmonary arterial pressure before and after ECCO2R treatment either in association with NIV or HNFCOT | Through study completion, an average of 2 years
  Echocardiographic measurement
Variation of tricuspid annluar plane systolic excursion before and after ECCO2R treatment either in association with NIV or HNFCOT | Through study completion, an average of 2 years
  Echocardiographic measurement
Variation of respiratory mechanic during ECCO2R+NIV | Through study completion, an average of 2 years
  Measurement of Respiratory Rate (breaths per minute)
Variation of dyspnea during ECCO2R+NIV | Through study completion, an average of 2 years
  Measurement of dyspnea through Borg dyspnea scale. (ranging from a minimum of 0 point, indicating no shortness of breath, to a maximum of 10 points, indicating maximum shortness of breath)
Variation of comfort during ECCO2R+NIV | Through study completion, an average of 2 years
  Measurement of comfort through Visual Analogic Scale for comfort, ranging from a minimum of 0 point, indicating no comfort, to a maximun of 10 point, indicating maximum comfort
Variation of respiratory mechanic during ECCO2R+HFNCOT | Through study completion, an average of 2 years
  Measurement of Respiratory Rate (breaths per minute)
Variation of dyspnea during ECCO2R+HFNCOT | Through study completion, an average of 2 years
  Measurement of dyspnea through Borg dyspnea scale, ranging from a minimum of 0 point, indicating no shortness of breath, to a maximum of 10 points, indicating maximum shortness of breath
Variation of comfort during ECCO2R+HFNCOT | Through study completion, an average of 2 years
  Measurement of comfort through Visual Analogic Scale for comfort, ranging from a minimum of 0 point, indicating no comfort, to a maximun of 10 point, indicating maximum comfort
Variation of breathing pattern during ECCO2R+NIV | Through study completion, an average of 2 years
  Measurement of expiratory tidal volume, expressed in mL
Variation of breathing pattern during ECCO2R+NIV | Through study completion, an average of 2 years
  Measurement of minute ventilation, expressed in liters/minute
Variation of acid-base balance during ECCO2R+NIV | Through study completion, an average of 2 years
  emogasanalysis
Variation of acid-base balance during ECCO2R+HFNCOT | Through study completion, an average of 2 years
  emogasanalysis

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Grasselli, Professor, Principal Investigator — Policlinico Hospital
Locations (1):
- Ospedale Maggiore Policlinico, Milan, Italy